CLINICAL TRIAL: NCT06419348
Title: 99mTc-QULIC-5-P1 SPECT Imaging in Patients With Prostate Cancer and Compared With 68Ga-PSMA-11 PET
Brief Title: 99mTc-QULIC-5-P1 SPECT Imaging in Patients With Prostate Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xiaoyang Zhang, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CYYY-KY-2023-268
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer Stage; PSMA; SPECT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 99mTc-QULIC-5-P1 (Experimental): Patients will receive a single administration of 99mTc-QULIC-5-P1
  Interventions: Drug: 99mTc-QULIC-5-P1

INTERVENTIONS:
Drug: 99mTc-QULIC-5-P1 — Each subject receives a single intravenous injection of 99mTc-QULIC-5-P1.

SUMMARY:
99mTc-QULIC-5-P1 is a new radiotracer targeting PSMA, which is promising as an excellent imaging agent applicable to PSMA positive prostate cancer. This study will investigate the safety, biodistribution and potential usefulness of 99mTc-QULIC-5-P1 SPECT imaging for the diagnosis of lesions in PSMA positive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Signed informed consent.
3. Patients with suspected or newly diagnosed or previously prostate cancer, with PSMA positive expression (supporting evidence may include MRI, CT, and pathology report, etc).

Exclusion Criteria:

1. Patients with PSMA negative expression.
2. Patients with pregnancy.
3. The inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.
4. Known or expected hypersensitivity to 99mTc-QULIC-5-P1 or any of its components.
5. Any serious medical condition or extenuating circumstance which the investigator feels may interfere with the procedures or evaluations of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | 15 days
  The sensitivity, specificity, and accuracy of 99mTc-QULIC-5-P1 SPECT

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No